CLINICAL TRIAL: NCT03034538
Title: An Open-Label Tolerability and Exploratory Efficacy Study of Zonisamide for Dyskinesias in Parkinson's Disease
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Site staffing
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-179
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Parkinson Disease; Parkinsonism; Dyskinesias
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Dyskinesias | interventions — Zonisamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 100mg (Active Comparator): Zonegran 100mg
  Interventions: Drug: Zonegran
- 200mg (Active Comparator): Zonegran 200mg
  Interventions: Drug: Zonegran

INTERVENTIONS:
Drug: Zonegran — 100mg
  Arms: 100mg
Drug: Zonegran — 200mg
  Arms: 200mg

SUMMARY:
In this 12-week, open-label pilot study, the investigators will enroll 20 subjects with Parkinson's Disease to determine if two doses of Zonisamide are tolerable and demonstrate clinical benefit for Dyskinesias. The primary outcome measure is tolerability, as determined by number of subjects able to complete the study on their originally assigned dosage. Secondary outcome measures will use the Unified Dyskinesia Rating Scale (UDysRS), comprised of an Objective Section and a Historical Section, to compare baseline to 6 and 12-week measurements. Additional analysis of the effect of Zonisamide on quality of life will be measured by the Parkinson's Disease Quality of Life Questionnaire (PDQ-39).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD
* Identified dyskinesias of the limbs or trunk as agreed upon by subject and investigator, with dyskinesias considered moderately to completely disabling (UPDRS question 33, greater or equal to 2)
* Able to provide informed consent and swallow capsules
* Stable doses of dopaminergic therapy for 2 weeks before and expected throughout the study.

Exclusion Criteria:

* Atypical parkinsonism
* Concurrent use of amantadine or active DBS where patient has some control over settings
* Prior surgery for PD
* Sulfa allergy or intolerance of zonisamide
* Significant concomitant medical illness in the opinion of the Principal Investigator (renal disease, liver disease)
* Pregnant subject or a subject who plans to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-04-08 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Unified Dyskinesia Rating Scale (UDysRS) | 12 weeks
  assesses involuntary movements encountered in the treatment of Parkinson's Disease. It consists of a Historical Section, divided into questionnaires about 1) on-dyskinesia and 2) off -dystonia, and an Objective Section, divided into 3) impairment and 4) disability scales. The Historical Section is scored from 0-60, and the Objective section is scored 0-44, where higher scores reflect greater difficulty or impairment.

SECONDARY OUTCOMES:
Parkinson's Disease Quality of Life Questionnaire (PDQ-39) | 12 weeks
  The 39-Item Parkinson's Disease Questionnaire (PDQ-39) is a commonly used measure of self-appraisal in PD.

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Health System, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No